CLINICAL TRIAL: NCT02499874
Title: Pharmacokinetics of EFV 400mg Once Daily During Pregnancy in HIV+ Women
Brief Title: SSAT063- Pharmacokinetics of Efavirenz 400 mg Once Daily During Pregnancy in HIV-1 Infected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Mylan Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT063
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: HIV
MeSH Terms: interventions — efavirenz; Tenofovir; Emtricitabine; Lamivudine; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single treatment arm (Experimental): All subjects will be administered oral Efavirenz 400mg together with the rest of the oral antiretroviral combination (tenofovir 245 mg/emtricitabine 200mg or tenofovir 245mg/lamivudine 300mg or lamivudine 300mg/zidovudine 600mg) throughout the study period
  Interventions: Drug: Efavirenz; Drug: tenofovir /emtricitabine; Drug: tenofovir/lamivudine; Drug: lamivudine/zidovudine

INTERVENTIONS:
Drug: Efavirenz — oral Efavirenz 400mg
  Other Names: Sustiva
Drug: tenofovir /emtricitabine — tenofovir 245 mg/emtricitabine 200mg
Drug: tenofovir/lamivudine — tenofovir 245mg/lamivudine 300mg
Drug: lamivudine/zidovudine — lamivudine 300mg/zidovudine 600mg

SUMMARY:
The purpose of the study is to measure the drug levels in your blood and to find out whether a reduced dose (400mg) of the anti-HIV medication Efavirenz is safe when taken during pregnancy.

The study will recruit HIV infected women who take Efavirenz as part of their anti-hiv treatment and who are pregnant.

Efavirenz has been shown to be safe in pregnancy and at the standard dose that everybody takes of 600mg once a day, it shows levels that are enough to treat HIV and give birth to a HIV negative baby.

Efavirenz at a dose of 400mg once daily works against HIV too but this dose has not been given to HIV positive pregnant women.

People with HIV may benefit from using a dose of efavirenz of 400mg instead of 600mg, as lower drug doses could have fewer side effects and be tolerated better.

Dose reduction would also make the drug cheaper. This would allow more people to be treated and free up money for other important work in the fight against HIV such as education and prevention programs.

However, it is not known whether 400mg of Efavirenz works as well as 600mg of Efavirenz during pregnancy and this is why the investigators are conducting this study, which aims to measure the amount of Efavirenz 400mg in HIV pregnant women's bodies when they are taking 400mg of Efavirenz once a day.

DETAILED DESCRIPTION:
Protocol Number: SSAT 063

EudraCT Number: 2014-002615-42

Name of Investigational Product: Sustiva

Name of active ingredients: Efavirenz

Study title:Pharmacokinetics of Efavirenz 400mg once daily during pregnancy in HIV-1 infected women

Name of Non Investigational Medicinal Product:

Two nucleoside reverse transcriptase inhibitors (tenofovir/ emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine)

Phase of study: Phase I

Objectives: The objectives of this study are:

* Primary

  -To investigate the pharmacokinetics of Efavirenz 400mg during pregnancy.
* Secondary

  * To investigate the safety and tolerability of Efavirenz 400mg during pregnancy.
  * To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure.

Study design: Two centre, approximately 18 weeks (excluding screening and follow up), open label, single treatment arm, pharmacokinetic study.

Indication: HIV in pregnancy

Methodology: Measurements of steady state pharmacokinetic profiles of efavirenz during the third trimester of pregnancy and 6 weeks postpartum in HIV-infected women on tenofovir/emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine plus Efavirenz 400mg once daily.

Planned sample size: The primary endpoint will be the comparison of efavirenz Ctrough during the third trimester of pregnancy versus postpartum. The efavirenz Ctrough from each patient will be compared between the two phases using geometric mean ratios (log10 transformed data). For this sequential design, a sample size of 25 patients would provide at least 80% power to detect a decrease in efavirenz Ctrough of 20% during the third trimester of pregnancy, compared to the postpartum phase.

Up to 35 individuals may be screened to achieve 25 women completing all PK phases.

Summary of eligibility criteria:

Pregnant HIV-infected women with:

* Undetectable viral load
* CD4 count > 100 cells/mm3
* Stable on tenofovir/emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine plus Efavirenz 600mg once daily for more than 12 weeks

Number of study centres: Two (London, UK and Kampala, Uganda)

Duration of treatment: Approximately 18 weeks: approximately four weeks prior to week 32 of pregnancy and up to 6 weeks postpartum (excluding screening and follow up visits)

Dose and route of administration: All subjects will be administered oral efavirenz 400mg together with the rest of the oral antiretroviral combination (tenofovir 245mg/emtricitabine 200mg or tenofovir 245mg/lamivudine 300mg or lamivudine 300mg/zidovudine 600mg) throughout the study period.

Criteria for evaluation: Pharmacokinetic parameters of efavirenz will be evaluated during the third trimester (gestational age week 32 +/- 3 weeks) and 6 weeks (+/- 4 weeks) postpartum.

Safety and tolerability of medications will also be assessed by questions, physical examination and laboratory parameters. These will be performed at regular intervals during the drug study.

At delivery, if possible, a cord blood sample will be taken and at the same time a blood sample from the mother will be taken.

Primary Endpoint:

Pharmacokinetics of efavirenz 400mg during pregnancy.

Secondary End point:

1. Safety and tolerability of efavirenz 400mg during pregnancy.
2. Association between genetic polymorphisms in drug disposition genes and drug exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. HIV-1-infected pregnant female, stable on two nucleos/tide analogues (tenofovir/emtricitabine or tenofovir/lamivudine or zidovudine/lamivudine) and efavirenz 600mg once daily for more than 12 weeks and willing to take efavirenz 400 mg once daily at gestational age of 28 weeks +/- 3 weeks.
3. Undetectable viral load (by local assay).
4. CD4 count > 100 cells/mm3.
5. Aged between 18 to 45 years, inclusive.

Exclusion Criteria:

1. Viral load ≥ 50 copies/mL (or detectable by local assay).
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations.
3. Positive blood screen for chronic hepatitis C (if available locally) or hepatitis B.
4. Current or recent (within 3 months) gastrointestinal disease.
5. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events.
6. Exposure to any investigational drug or placebo within 3 months prior to first dose of study drug.
7. Use of any other drugs, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-08; Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC and Ctrough) of Efavirenz 400mg during pregnancy and postpartum. | 24 weeks
  The pharmacokinetic parameters calculated for efavirenz will be trough concentration (Ctrough), defined as the concentration at 24 hours after the observed drug dose, the maximum observed plasma concentration (Cmax), elimination half-life (t1/2), time point at Cmax (Tmax), and total drug exposure, expressed as the area under the plasma concentration-time curve from 0-24 hours after dosing (AUC0-24h). Efavirenz pharmacokinetic parameters measure during the third trimester of pregnancy and postpartum will be compared by calculating geometric mean ratios and 90% confidence intervals.

SECONDARY OUTCOMES:
Safety and tolerability (based on physical examination, laboratory tests and the DIVISION OF AIDS (DAIDS) table for granding the severity of adult and and the pediatric adverse events of Efavirenz 400mg during pregnancy and postpartum | 24 weeks
  Safety and tolerability of medications will also be assessed by questions, physical examination and laboratory parameters. These will be performed at regular intervals during the drug study.
Association between polymorphisms in drug disposition genes and exposure in order to understand whether polymorphism of certain genes encoding for efavirenz metabolic enzymes are behind differences in efavirenz pharmacokinetics between people | 24 weeks
  candidate gene approach will be utilised to examine loci of interest. This procedure will provide potentially important information on genetic influences on plasma drug concentrations and give insight into how to improve the management of HIV-infected patients by individualising therapy. These studies will not be powered for genetic associations but will enable us to build a data base of genotype-phenotype. Prospective genetic studies would need to be planned based on these preliminary data.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, MBBS,MD,PhD, Principal Investigator — St. Stephen's AIDS Trust; Mohammed Lamorde, MBBS, Principal Investigator — Infectious Diseases Institute (IDI)
Locations (1):
- St Stephen's Centre, Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNAIDS is the leading advocate for worldwide action against HIV/AIDS. It promotes partnerships among and between other UN agencies, governments, corporations, media, sports and religious organizations, community-based groups — http://www.unaids.org
- See also: BHIVA (the British HIV Association) is an organisation that represents healthcare professionals working in HIV in the UK. Its guidelines set out the medical and other care people living with HIV can expect to receive in the UK — http://www.bhiva.org